CLINICAL TRIAL: NCT06850636
Title: Higher vs Lower Lumber Epidural Catheter Insertion During Labour: A Randomised Trial to Compare Efficacy.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Rotunda Hospital (Other)
Responsible Party: Principal Investigator, Tom Drew, Principal Investigator and Consultant Anaesthesiologist, The Rotunda Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC-2024-027
Record Dates: First submitted 2025-02-18; First posted 2025-02-27 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Labour Analgesia, Epidural Anaesthesia
MeSH Terms: interventions — Analgesia, Epidural

STUDY DESIGN:
Intervention Model Description: This is a prospective randomised study where women will be randomised to a high or low epidural catheter to determine which is superior for maternal analgesia efficacy and satisfaction.
  Randomised to intervention 'high epidural' or 'low epidural' groups. Within these groups there are two subgroups based on the specific lumbar vertebral level; high epidural (L 1,2 or L 2,3 levels) and low epidural (L 3,4 or L 4,5 levels).
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Epidural analgesia performed at a higher lumbar epidural level (Active Comparator): Epidural analgesia performed using Programmed Intermittent Epidural Boluses using an epidural catheter at a higher lumbar epidural level sited at L1,L2 or L2,L3
  Interventions: Procedure: Epidural Analgesia
- Epidural analgesia performed at a lower lumbar epidural level (Active Comparator): Epidural analgesia performed using Programmed Intermittent Epidural Boluses using an epidural catheter sited at lower epidural level (L3,L4 or L4,L5)
  Interventions: Procedure: Epidural Analgesia

INTERVENTIONS:
Procedure: Epidural Analgesia — Labour epidural analgesia

SUMMARY:
This study will randomise pregnant women to labour epidural at a higher versus a lower lumbar level. Outcomes relating to success or failure of the epidural catheter at this level will be assessed.

DETAILED DESCRIPTION:
Epidural analgesia is widely used in different types of surgeries and procedures. Pregnant women in labour compromise the single largest group benefiting from epidural analgesia. During first stage of labour (dilatation of the cervix), an epidural should cover the sensory dermatomes from T10 to L1 to achieve a good pain relief. In the second stage of labour (descent of the baby through the cervical canal), pain is mediated via S2-S4 nerve roots. Accordingly, labour epidurals are commonly placed at the lower lumbar (L3-L4) interspace.1 A study was conducted by Moore et al., comparing high vs low lumbar epidural, showed that lower epidurals provide superior perineal analgesia, when used with a patient-controlled epidural analgesia (PCEA) infusion with continuous epidural infusion (CEI), but provided less pain relief early in labour. Another study, a metanalysis showed that another mode of delivery of the local anaesthetics is more effective; which is the Programmed Intermittent Epidural Boluses (PIEB) with PCEA. The incidence of breakthrough pain, the rates of local anaesthetic usage were significantly reduced, the labour duration was statistically shorter, and the maternal satisfaction score was significantly improved in the PIEB + PCEA group compared with that in the CEI + PCEA group.

This is a prospective randomised study where women will be randomised to a high or low epidural catheter to determine which is superior for maternal analgesia efficacy and satisfaction.

Randomised to intervention 'high epidural' or 'low epidural' groups. Within these groups there are two subgroups based on the specific lumbar vertebral level; high epidural (L 1,2 or L 2,3 levels) and low epidural (L 3,4 or L 4,5 levels).

ELIGIBILITY:
Inclusion Criteria:

Women electing to have epidural analgesia in labour

Exclusion Criteria:

Known contraindication to epidural analgesia. Neurological illness Multiple gestation Fetal abnormalities In distress or requiring immediate epidural catheter placement

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Composite outcome: Failure of Labour epidural catheter or PIEB protocol | During labour
  Composite outcome of 1/Failure to insert labour epidural at the assigned level OR 2/ Labour epidural catheter requires resiting OR 3/ Healthcare worker top up due to pain OR 4/ Failure of epidural conversion to epidural anaesthesia if caesarean section required

SECONDARY OUTCOMES:
Pain score | 60 minutes post delivery and at postnatal follow up.
  Pain scores taken 60 minutes after insertion of epidural catheter and retrospective pain scores assessed during second stage of labour taken at follow up visit. Pain scores to be assessed using a visual analogue score of 0-10, where 0 is no pain at all and 10 is the worst pain.
Dermatomal sensory level assessed using cold sensation | 60 minutes after insertion of the epidural catheter
  Dermatomal sensory level assessed 60 minutes after insertion of the epidural catheter using ice. Assessed by placing ice at the L1 dermatome, and move cranially or caudally until the patient notices a change in cold sensation.
Bromage score | 60 minutes after insertion of labour epidural catheter
  Motor block assessed at 60 minutes
Patient Satisfaction | At follow up visit within 24 hours
  Patient satisfaction assessed at follow up visit, assessed using a scale of 0-10 where 0 is extremely dissatisfied and 10 is extremely satisfied.
Depth of the epidural space | At time of insertion
  The depth to the epidural space in cm
Difficulty of epidural insertion | At time of epidural insertion
  Difficulty of epidural insertion as perceived by the clinican, on a scale on 1-4 where 1 is easy and 4 is very difficult.

CONTACTS AND LOCATIONS:
Locations (1):
- The Rotunda Hospital, Dublin, Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No